CLINICAL TRIAL: NCT04924140
Title: A Randomized, Open-Label, Parallel-Arm Study to Assess the Absolute Bioavailability of a Single, Fixed Subcutaneous Dose of Aducanumab (BIIB037) Compared to a Single, Weight-Based Intravenous Dose in Healthy Volunteers
Brief Title: A Study to Assess Absolute Bioavailability of Aducanumab in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 221HV103
Record Dates: First submitted 2021-06-08; First posted 2021-06-11 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — aducanumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aducanumab Intravenous (Experimental): Participants will receive aducanumab as body weight-based dose, via IV infusion for approximately 1 hour on Day 1.
  Interventions: Drug: Aducanumab
- Aducanumab Subcutaneous (Experimental): Participants will receive aducanumab as fixed dose, via SC injection on Day 1.
  Interventions: Drug: Aducanumab

INTERVENTIONS:
Drug: Aducanumab — Administered as specified in the treatment arm
  Other Names: BIIB037

SUMMARY:
The primary objective of this study is to evaluate the absolute bioavailability of a single, fixed subcutaneous (SC) dose of aducanumab compared with a single weight-based intravenous (IV) dose of aducanumab in healthy volunteers.

The secondary objectives of this study are to assess the safety and tolerability of aducanumab administered SC in healthy volunteers and to characterize additional pharmacokinetic (PK) parameters of a single, fixed SC dose of aducanumab and a weight-based IV dose of aducanumab in healthy volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a body mass index (BMI) between 18 and 30 kilograms per meter square (kg/m^2), inclusive.
* Have a negative test result for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) on Day -1.

Key Exclusion Criteria:

* History of any clinically significant cardiac, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease, or other major disease, as determined by the investigator.
* History of severe allergic, anaphylactic, or systemic hypersensitivity reactions, or of any allergic reactions that in the opinion of the investigator are likely to be exacerbated by aducanumab, the excipients contained in the formulation, and if appropriate, and diagnostic agents to be administered during the study.
* Chronic, recurrent, or serious infection (e.g., pneumonia, septicemia), as determined by the investigator, within 90 days prior to screening or between screening and Day -1.
* Any immunization or vaccination given within 10 days prior to Day 1 and for 10 days after Day 1.
* Current enrollment in any other drug, biological, device, or clinical study, or treatment with an investigational drug or approved therapy for investigational use within 30 days prior to Day -1, or 5 half-lives, whichever is longer.
* Prior exposure to the study treatment or previous participation in this study or previous studies with aducanumab.
* Mini mental state examination (MMSE) score of <27 at screening.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUCinf) of Aducanumab | Up to Day 85
Maximum Observed Concentration (Cmax) of Aducanumab | Up to Day 85

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Day 85
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose results in death; in the view of the investigator, places the participant at immediate risk of death (a life-threatening event); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect or is a medically important event.
Number of Participants with Clinically Significant Abnormalities in Vital Signs | Up to Day 85
Number of Participants with Clinically Significant Abnormalities in 12-Lead Electrocardiograms (ECGs) | Up to Day 85
Number of Participants with Clinically Significant Abnormalities in Laboratory Assessments | Up to Day 85
Area Under the Concentration-Time Curve from Time 0 to Time of the Last Measurable Concentration (AUClast) of Aducanumab | Up to Day 85
Time to Reach Maximum Observed Concentration (Tmax) for Aducanumab Administered SC | Up to Day 85
Elimination Half-Life (t½) of Aducanumab | Up to Day 85
Volume of Distribution (Vd) or Apparent Volume of Distribution (V/F) of Aducanumab | Up to Day 85
Clearance (CL) or Apparent Clearance (CL/F) of Aducanumab | Up to Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (2):
- United States (2):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Qps-Mra, Llc, South Miami, Florida

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/